CLINICAL TRIAL: NCT03327285
Title: A Study Evaluating Safety and Efficacy of CBM.CD19-targeted Chimeric Antigen Receptor T Cells (C-CAR011) Treatment in Subjects With Acute Lymphoblastic Leukemia(ALL) After Hematopoietic Stem Cell Transplantation（HSCT）
Brief Title: C-CAR011 Treatment in Subjects With ALL After HSCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Peking University People's Hospital (Other)
Collaborators: Shanghai AbelZeta Ltd. (Industry)
Responsible Party: Principal Investigator, Xiaojun Huang,MD, Chair, Peking University People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017PHB033-01; CBMG-C2017004 (Other: CBMG)
Record Dates: First submitted 2017-08-17; First posted 2017-10-31 (Actual); Last update posted 2020-10-01 (Actual); Status verified 2020-09

CONDITIONS: Acute Lymphoblastic Leukemia(ALL)
Keywords: Acute lymphoblastic leukemia; Hematopoietic stem cell transplantation; Anti-CD19 chimeric antigen receptor T-cell
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- C-CAR011 (Experimental): The amount of cells received：1.0-5.0×10^6 CAR+T cells/kg
  Interventions: Biological: C-CAR011

INTERVENTIONS:
Biological: C-CAR011 — CBM.CD19-targeted chimeric antigen receptor T cells(C-CAR011)
  Other Names: Anti-CD19 chimeric antigen receptor T cells (C-CAR011)

SUMMARY:
This is a single-center, prospective clinical study evaluating safety and efficacy of C-CAR011 treatment in subjects with ALL after HSCT

DETAILED DESCRIPTION:
A study evaluating safety and efficacy of CBM.CD19-targeted chimeric antigen receptor T cells (C-CAR011) treatment in subjects with acute lymphoblastic leukemia(ALL) after hematopoietic stem cell transplantation（HSCT）. The amount of cells received：1.0-5.0×10^6CAR+T cells/kg

ELIGIBILITY:
Inclusion Criteria:

* Age 15-65 years old, male or female.
* Volunteered to participate in this study and signed informed consent.
* Meet the two populations above.
* Histologically diagnosed as CD19+B-ALL.
* 100% T lymphocytes of donor.
* Treatment without chemotherapy and antibody therapy within 2 weeks prior to C-CAR011 therapy.
* Left ventricular ejection fraction (LVEF) ≧ 50%, no evidence of pericardial effusion and clinically significant arrhythmias.
* Baseline oxygen saturation ≧ 92% on room air and with normal pulmonary function, no evidence of active lung infection.
* Expected survival ≧ 3 months.
* Eastern cooperative oncology group (ECOG) performance status of 0 or 1.

Exclusion Criteria:

* History of allergy to cellular products.
* Any kind of these laboratory testing: serum total bilirubin≧2.0mg/dl, serum albumin<35g/L, ALT, AST≧3×ULN, serum creatinine≧2.0mg/ dl,platelets<20×109/L.
* The subjects had active aGVHD with II-IV degrees (Glucksberg degrees) or active moderate to severe cGVHD.
* Severe uncontrolled infection (mycotic, bacterial, virus and so on).
* Any central nervous system leukemia(CNS2, CNS3) , with insensitive to intrathecal injection of or radiotherapy of head/spine; but effectively controlled cases will be eligible.
* The subjects were treated CART cells or DLI after HSCT.
* Bone marrow failure syndrome（BMF） after allogeneic hematopoietic stem cell transplantation.
* Any genetically modified T cell therapy.
* History of heavy drinking, drug taking or mental disease.
* Participated in any other clinical trial within one month prior to enrollment.
* Women who are pregnant or lactating or have breeding intent in 6 months.
* The investigators believe that any increase in the risk of the subject or interference with the results of the trial.

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2021-02-28 (Estimated); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
TEAEs | 2 months
  TEAEs evaluated after C-CAR011 infusion
GVHD | 2 months
  GVHD evaluated after C-CAR011 infusion

SECONDARY OUTCOMES:
Recurrence rate | 6 and 12 months
  Recurrence rate
OS | 12 months
  Overall survival (OS) after C-CAR011 infusion
PFS | 12 months
  Progression free survival（PFS）after C-CAR011 infusion
Remission rate | 2 weeks to 3 months
  MRD negative after C-CAR011 infusion

CONTACTS AND LOCATIONS:
Overall Officials: Xiaojun Huang, Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University Institute of Hematology, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided